CLINICAL TRIAL: NCT00010374
Title: Multi-Center Pivotal Study of NeuRx RA/4 Ventilatory Assist Device
Brief Title: Electrical Activation of The Diaphragm for Ventilatory Assist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); Shepherd Center, Atlanta GA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-0000-0009
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injury; Quadriplegia
Keywords: Diaphragm for Ventilatory Assist; environmental/toxic disorders; neurologic and psychiatric disorders; rare disease; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Neurologic Manifestations; Mental Disorders; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeuRx DPS (Experimental): Laparoscopic implantation of 4 NeuRx DPS electrodes and subsequent pacing using the DPS system.
  Interventions: Device: NeuRx DPS

INTERVENTIONS:
Device: NeuRx DPS — Laparoscopic implantation of diaphragm electrodes and subsequent pacing with the NeuRx DPS.

SUMMARY:
OBJECTIVES:

The objectives of this study are to test the Diaphragm Pacing Stimulation (DPS) System for treating chronic ventilatory insufficiency in persons with respiratory muscle paralysis. The hypothesis being tested in the clinical trial is that laparoscopic stimulation of the diaphragm at the motor point with intramuscular electrodes is safe and effective in providing significant ventilatory support to individuals who are otherwise dependant on a mechanical ventilator. Patients in our initial study group have all suffered from high-level spinal cord injury and were full-time dependant on positive pressure mechanical ventilation prior to inclusion.

DETAILED DESCRIPTION:
System: NeuRx RA/4 Diaphragm Pacing Stimulation System

Summary:

The NeuRx-RA/4 is intended to be used by individuals that have sustained a spinal cord injury, requiring aid with respiration. The device connects to the diaphragm which delivers current to stimulate muscle contractions to aid in respirations.

This device currently holds an Investigational Device Exemption No. G920162 in the United States and is currently undergoing clinical trials at University Hospitals (Cleveland), Shepherd Center (Atlanta) and Vancouver (Canada).

Introduction:

The purpose of the study is to determine if a new, investigational diaphragm pacing system can provide part or full time respiratory support to spinal cord injured persons who normally need a mechanical ventilator. Patients with high-level spinal cord injuries typically experience chronic ventilatory insufficiency due to respiratory muscle paralysis; these patients must be supported predominantly through positive pressure mechanical ventilation with a ventilator.

The diaphragm pacing system (NeuRx-RA/4) provides an electrical signal to the motor point of the muscle that causes the diaphragm to contract and allows patients to breathe more naturally.

Synapse Biomedical, in conjunction with Case Western Reserve University and University Hospitals of Cleveland, are evaluating activating the diaphragm with percutaneous intramuscular electrodes implanted laparoscopically. This eliminates any direct contact with the phrenic nerve, allows all circuitry and electronics to remain outside the body, and provides direct, selective activation to each hemidiaphragm.

The NeuRx RA/4 Diaphragm Pacing Stimulation (DPS) System has been implanted in 49 individuals with high-level spinal cord injury, resulting in over 20 years of cumulative active implantation time. The longest term patient was implanted March 6, 2000 and has been using the DPS System as his sole means of respiratory support for over five years. With the exception of the second patient, who does not meet our revised inclusion criteria and has gained no benefit from the implant, all of the remaining patients have been able to achieve significant tidal volumes with the DPS System. Based on the current results, the NeuRx RA/4 DPS System has demonstrated safety and efficacy in patients with high-level spinal cord injury.

Given the results to date the study has demonstrated preliminary efficacy in this patient population. With no unexpected significant adverse events reported the NeuRx RA/4 DPS System has performed reliably and safely in this patient population.

Device Description: The NeuRx RA/4 Respiratory System is manufactured by Synapse Biomedical. The NeuRx RA/4 System comprises the following components: an external, battery powered Stimulator Device, an associated Programmer/Controller, Intramuscular Electrodes, associated percutaneous Lead Wires, a Surgical Placement Tool Set, and a surgical Mapping Station.

Inclusion Criteria:

* Age 18 years or older
* Cervical spinal cord injury dependent on mechanical ventilation
* Clinically stable following acute spinal cord injury
* Bilateral phrenic nerve function clinically acceptable as demonstrated with EMG recordings and nerve conduction times
* Diaphragm movement with stimulation visible under fluoroscopy
* Clinically acceptable oxygenation on room air (>90%)
* Hemodynamically stable
* No medical co-morbidities that would interfere with the proper placement or function of the device
* Committed primary caregiver
* Negative pregnancy test in females of child-bearing potential
* Informed consent from patient or designated representative

Exclusion Criteria:

* Co-morbid medical conditions that preclude surgery
* Active lung disease (obstructive, restrictive or membrane diseases)
* Active cardiovascular disease
* Active brain disease
* Hemodynamic instability or low oxygen levels on room air
* Hospitalization for or a treated active infection within the last 3 months
* Significant scoliosis or chest deformity
* Marked obesity
* Anticipated poor compliance with protocol by either patient or primary caregiver.
* Currently breastfeeding

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cervical spinal cord injury dependent on mechanical ventilation
* Clinically stable following acute spinal cord injury
* Bilateral phrenic nerve function clinically acceptable as demonstrated with EMG recordings and nerve conduction times
* Diaphragm movement with stimulation visible under fluoroscopy
* Clinically acceptable oxygenation on room air (>90%)
* Hemodynamically stable
* No medical co-morbidities that would interfere with the proper placement or function of the device
* Committed primary caregiver
* Negative pregnancy test in females of child-bearing potential
* Informed consent from patient or designated representative

Exclusion Criteria:

* Co-morbid medical conditions that preclude surgery
* Active lung disease (obstructive, restrictive or membrane diseases)
* Active cardiovascular disease
* Active brain disease
* Hemodynamic instability or low oxygen levels on room air
* Hospitalization for or a treated active infection within the last 3 months
* Significant scoliosis or chest deformity
* Marked obesity
* Anticipated poor compliance with protocol by either patient or primary caregiver
* Currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Onders, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (5):
- United States (4):
  - Craig Hospital, Englewood, Colorado
  - Shepherd Center, Atlanta, Georgia
  - University Hospital Of Cleveland, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
- Vancouver CoastHealth, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients who have suffered from high-level spinal cord injury, are full-time dependent on positive pressure mechanical ventilation and have intact bilateral phrenic nerves.
Pre-assignment Details: One participant had a false positive phrenic nerve test after consent
Groups:
- Treatment: Laparoscopic implantation of 4 NeuRx DPS electrodes and subsequent pacing using the DPS system.
Period: Overall Study
Arm/Group | Treatment
Started | 54
Completed | 53 (One compassionate use participant was withheld from analysis per FDA instructions)
Not Completed | 1
Not completed — False positive phrenic nerve test | 1

BASELINE CHARACTERISTICS:
Population: Patients with stable, high spinal cord injuries with stimulatable diaphragms, but lack control of their diaphragms that were implanted with the NeuRx DPS electrodes and able to condition their diaphragm using the study device.
Groups:
- NeuRx DPS: Laparoscopic implantation of 4 NeuRx DPS electrodes and subsequent pacing using the DPS system.
  NeuRx DPS: Laparoscopic implantation of diprapagm electrode and subsequent pacing with the NeuRx DPS.
Arm/Group | NeuRx DPS
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 41
Region of Enrollment [Number; unit: participants]
  Canada | 1
  United States | 50
  Iceland | 2
Time since injury [Mean (Standard Deviation); unit: years] | 5.425 (6.75)

OUTCOME MEASURES:

1. Primary Outcome: Enrolled Subjects Achieve Clinically Acceptable Tidal Volume Sustained Over a Continuous 4 Hour Period.
Description: Number of enrolled subjects that successfully maintained clinically acceptable tidal volumes greater than basal requirements over a continuous 4 hour period.
Time Frame: Within one year after implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants
  Success: Vt>Basal Req. Continuous use > 4 hours | 52
  Partial success: Vt>Basal Req. max use < 4 hours | 1
Statistical Analysis 1: Comparison: Treatment; Test type: Other — Performance goal of 35%; p < 0.001, Exact two-sided binomial test; Exact two-sided binomial test = 96.2, 95% CI 2-sided [87.0 to 99.5]

2. Secondary Outcome: Achieve Clinically Acceptable Basal Metabolic Requirement of Tidal Volume Measured in ml During Chronic Stimulation.
Description: To evaluate the ability of NeuRx DPS therapy to replace mechanical ventilation for patients on a chronic use basis, a secondary indicator of this objective is tidal volume (Vt) measured in ml during chronic stimulation.
Time Frame: Within one year after implantation
Population: Participants with high level spinal cord injury that are dependent on mechanical ventilation and have intact phrenic nerves.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- NeuRx Implanted Patients: SCI patients who received NeuRx DPS implants
Arm/Group | NeuRx Implanted Patients
Number analyzed (Participants) | 53
ml | 745.6 (217.7)

3. Secondary Outcome: Number of Patients That Use NeuRx DPS to Breathe Without the Assistance of a Mechanical Ventilator for 24 Continuous Hours a Day
Description: Number of patients that can achieve at least 24 hours daily use of the NeuRx DPS without the assistance of a mechanical ventilator.
Time Frame: Within one year of implantation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NeuRx Implanted Patients
Number analyzed (Participants) | 53
Participants | 31

ADVERSE EVENTS:
Time Frame: 1 year from date of enrollment
Description: No details to include
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 4/53
Serious Adverse Events (participants affected / at risk) | 8/53
Other Adverse Events (participants affected / at risk) | 38/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=53)
Death while device was not in use (General disorders) | 2 (2) — Two of the deaths occurred while the patient was being mechanically ventilated and not paced. In one case the patient was found lifeless during the night; in another case the patient died of cardiac arrhythmia and subsequent cardiac failure.
Death while device was in use (General disorders) | 2 (2) — One patient was observed to lose consciousness while the device was functioning. A second patient died of septic shock due to urosepsis and was using the device prior to a hypotensive arrest. No device malfunction was observed.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (10)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2)
Acute Polynephritis (Renal and urinary disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (2)
Chest Pain (Cardiac disorders) | 1 (1)
Elevated Temperature (Infections and infestations) | 2 (2)
Blood from and around treacheostomy tube (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=53)
Urinary tract infection (Renal and urinary disorders) | 6 (10)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain/discomfort with stimulation (Musculoskeletal and connective tissue disorders) | 3 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (11) — without evidence of respiratory distress, hypoxemia or aspiration
Increased secretions (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Low oxygen saturation/tidal volume (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Capnothorax (Respiratory, thoracic and mediastinal disorders) | 21 (21)
Broken External Wire (Product Issues) | 7 (12)
External Equipment Failure (Product Issues) | 8 (10)
Elevated Temperature (General disorders) | 3 (6)
Broken Anode (Product Issues) | 6 (8)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 (9) — Includes Cold/Nasal Congestion
Pressure Sore (Skin and subcutaneous tissue disorders) | 3 (4)
Pain/Discomfort no device use (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No